CLINICAL TRIAL: NCT06144385
Title: A Phase 1, Single-arm, Open-label, Dose-escalation Study of JWATM204 as T Cell-targeted Immunotherapy in the Treatment Amongst Subjects With Advanced Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Ming Ju Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JWATM204001
Record Dates: First submitted 2023-11-15; First posted 2023-11-22 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Liver Carcinoma; Hepatic Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-GPC3 T cells (Experimental): The safety and efficacy of JWATM204 will be evaluated in a Bayesian Optimal Interval Design (BOIN) dose escalation approach. 3 CAR-T dose levels will be tested in this study: 1×10^8, 3×10^8, 10×10^8, and 30×10^8 CAR-T cells will be explored.
  Interventions: Biological: CAR-GPC3 T cells

INTERVENTIONS:
Biological: CAR-GPC3 T cells — Subjects will undergo leukapheresis to isolate peripheral blood mononuclear cells (PBMCs) for the production of JWATM204 . During JWATM204 production, subjects will receive a preconditioning chemotherapy regimen of cyclophosphamide and fludarabine to deplete the lymphocytes. After lymphodepletion, subjects will receive single-dose treatment with JWATM204 by intravenous (IV) injection.
  Other Names: JWCAR204

SUMMARY:
This is a single arm, open-label, dose escalation clinical study to evaluate the safety and efficacy of infused autologous GPC3-directed CAR-T in patients with advanced hepatocellular carcinoma refractory to prior systematic treatments.

ELIGIBILITY:
Inclusion Criteria:

1. 18-75 years-old, male or female
2. Voluntarily willing to participate in the study and sign the written informed consent form
3. Life expectation ≥12 weeks
4. Eastern Cooperative Oncology Group (ECOG) performance status scale ≤1
5. Histologically-confirmed hepatocellular carcinoma (HCC)
6. No benefits from curative surgery or other local therapies are expected at screening, judged by investigators
7. Radiologically-confirmed progression disease after at least one prior line of systematic treatment and limited benefits from current available options for hepatocellular carcinoma are expected at screening, judged by investigators
8. Fresh samples or formalin-fixed paraffin-embedded (FFPE) samples, immunohistochemistry (IHC)-stained GPC-3 positive
9. Per RECIST v1.1, at least one measurable lesion
10. Barcelona Clinic Liver Cancer (BCLC) stage C or B and Child-Pugh ≤7
11. No active infections of hepatitis B virus
12. Adequate organ functions
13. Adequate venous access for apheresis
14. Non-hematological AEs induced by previous treatment must have recovered to CTCAE ≤1, except for alopecia and peripheral neuropathy
15. Women of childbearing potential must agree to use an effective and reliable contraceptive method during 28 days prior to lymphodepletion to 1 year post infusion; Male patients who have not undergone vasectomy and have sexual activity with women of childbearing potential must agree to the use of a barrier contraceptive method since lymphodepletion to 1year post infusion, and sperm donation is prohibited during the study
16. Women of childbearing potential must have negative serum β-human chorionic gonadotropin (β-hCG) test result at screening and 48 hours prior to lymphodepletion

Exclusion Criteria:

1. Active brain metastasis
2. Primary lesion or infused lesions with the longest diameter ≥15 cm, or other potential risk which might not be appropriate for further study treatment judged by the investigator
3. Another primary malignancy within 3 years (with some exceptions for completely-resected early-stage tumors)
4. Systematic autoimmune disorders requiring long-term systematic immunosuppression
5. Previously treated with any genetically engineered modified T-cell therapy nor other cell-gene therapy
6. Active infections of hepatitis C virus (HCV), human immunodeficiency virus (HIV), or syphilis
7. Uncontrolled or active infection at screening, prior to apheresis, 72 hours prior to lymphodepletion or 5 days prior to JWATM204 infusion
8. With severe cardiovascular disease History or presence of clinically-relevant central nervous system (CNS) disorders
9. With clinically-significant CNS disorders
10. Current presence of or previously with hepatic encephalopathy
11. ≥G2 hemorrhage within 30 days prior to screening, or in need of long-term anticoagulants
12. Pregnant or lactating women
13. Not satisfying pre-defined wash-out period for apheresis
14. Received plasma exchange within 14 days prior to apheresis
15. Unable or unwilling to comply with the study protocol, judged by the investigator, or other situations implying that the subject might not be appropriate to participate in the study
16. Vaccinated with live vaccinations against infectious diseases within 8 weeks prior to JWATM204 infusion
17. Previously allergic or intolerable to JWATM204 or its components

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-03-24 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Rate of dose-limiting toxicities (DLTs) | 28 days
  Dose-limiting toxicity (DLT) is defined as an adverse event that occurred within 28 days after JWATM204 infusion that met any of the following criteria. Any grade ≥3 nonhematologic toxicity associated with JWATM204 that has not resolved to ≤ grade 2 within 7 days, excluding clinically insignificant abnormalities in laboratory indicators Hematologic toxicity Grade ≥3 anaphylaxis Grade ≥3 infection did not resolve to grade ≤2 within 7 days after anti-infective treatment. ≥ grade 3 autoimmune toxicity during treatment Grade ≥3 cytokine release syndrome (CRS) during treatment that did not resolve to grade ≤2 within 72 hours. Grade ≥3 CAR-T cell-associated encephalopathy syndrome/immune effector cell-associated neurotoxicity syndrome (CRES/ICANS) that did not resolve to grade ≤2 within 72 hours. Grade 5 events of any nonmalignant cause.
Rate and severity of adverse events (AEs) and severe adverse events (SAEs) | 2 years
  An AE is defined as any unfavorable and unintended sign, symptom, or disease (new or worsening) temporally associated with the use of study therapy, regardless of whether or not a causal relationship with the study therapy can be determined.
Rate and severity of clinically-significant abnormalities in laboratory testings | 2 years
  Clinically-significant abnormalities in laboratory testings.

SECONDARY OUTCOMES:
Copy number of the vector transgene of JWATM204 in peripheral blood | 1 year
  The pharmacokinetic parameters of JWATM204 will be evaluated by quantitative polymerase chain reaction (qPCR) for the copy number of the vector transgene of JWATM204 in peripheral blood to evaluate T-cell expansion and persistence.
Objective response rate (ORR) | 2 years
  Proportion of patients whose tumor volume has reached a predetermined value and can maintain a minimum time limit, including complete response and partial response patients.
Disease Control Rate (DCR) | 2 years
  The percentage of patients with advanced or metastatic cancer who have achieved complete response, partial response and stable disease to a therapeutic intervention in clinical trials of anticancer agents.
Progression-free survival (PFS) | 2 years
  Defined as time from randomisation to first progression by investigator assessment using revised Response Evaluation Criteria in Solid Tumours (RECIST) guidelines (version 1.1) or death (by any cause in the absence of progression)
Overal survival (OS) | 2 years
  Defined as the time from randomisation to death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Tao Zhang, MD, PhD, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Tao Zhang, Wuhan, Hubei, China